CLINICAL TRIAL: NCT00534170
Title: Randomized Controlled Field Trial of a Probiotics to Assess Its Role in The Prevention of Acute Diarrhoeal Diseases in Children
Brief Title: Randomized Controlled Field Trial of a Probiotics to Assess Its Role in Preventig Diarrhoea
Acronym: Yakult
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indian Council of Medical Research (Other Government)
Collaborators: Yakult Honsha Co., LTD (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YH-001 NICED 010
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-06

CONDITIONS: Diarrhea
Keywords: Probiotic; Prevention of diarrhoea; Nutritional status
MeSH Terms: conditions — Diarrhea | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A,F,T,K (Experimental): Two arms are for intervention and two are for control or placebo
  Interventions: Dietary Supplement: Probiotic (Yakult)

INTERVENTIONS:
Dietary Supplement: Probiotic (Yakult) — It is a dietary supplement ,65 ml containing 15 billion lactobacillus
  Other Names: Yakult

SUMMARY:
A therapeutic as well as preventive role of probiotics has been suggested from results of different studies using different probiotics that have been tested, usually lactic acid producing bacteria such as lactobacillus, bifidobacterium and streptococcus species. The supplementation of probiotics to infants may also have a prophylactic effect against acute diarrhoeal diseases.

In the present proposal, we plan to examine if daily intake of a probiotic beverage, which includes 15 billion probiotic Lactobacilli, has a beneficial role in protecting children from infectious diarrhea in Kolkata.

OBJECTIVES

Primary objectives:

1. To assess the impact of probiotics in the prevention of acute diarrhoeal diseases in children
2. To assess the impact of probiotics on nutrition and growth of the children

Secondary Objectives:

1. Reduction in duration, frequency of diarrhoea
2. Identification of pathogens causing diarrhoea
3. Examination of faecal microflora

STUDY DESIGN

It will be a double blind randomized controlled field trial involving 4000 children aged between 1 and 5 years in an urban slum of Kolkata, India. The 4000 children will be identified through demographic survey. The study will be double blinded where the study arm will receive Probiotic drink, which includes 15 billion probiotic Lactobacilli, one bottle (65ml) daily (under supervision of a Health Worker) for 12 weeks and the control arm will receive a similar drink without the lactobacilli (Nutrient drink) daily for 12 weeks. Randomization will be done in a ratio of 1:1, i.e., the study arm and control arm will include 2000 children each. All the children under the study will be visited daily by a health worker who will supervise intake of Probiotic drink or Nutrient drink by the children. All the children will be followed up daily for 24weeks for identification of acute diarrhoea cases.

DETAILED DESCRIPTION:
A therapeutic as well as preventive role of probiotics has been suggested from results of different studies using different probiotics that have been tested, usually lactic acid producing bacteria such as lactobacillus, bifidobacterium and streptococcus species. The supplementation of probiotics to infants may also have a prophylactic effect against acute diarrhoeal diseases.

In the present proposal, we plan to examine if daily intake of a probiotic beverage, which includes 15 billion probiotic Lactobacilli, has a beneficial role in protecting children from infectious diarrhea in Kolkata.

OBJECTIVES

Primary objectives:

1. To assess the impact of probiotics in the prevention of acute diarrhoeal diseases in children
2. To assess the impact of probiotics on nutrition and growth of the children

Secondary Objectives:

1. Reduction in duration, frequency of diarrhoea
2. Identification of pathogens causing diarrhoea
3. Examination of faecal microflora

STUDY DESIGN

It will be a double blind randomized controlled field trial involving 4000 children aged between 1 and 5 years in an urban slum of Kolkata, India. The 4000 children will be identified through demographic survey. The study will be double blinded where the study arm will receive Probiotic drink, which includes 15 billion probiotic Lactobacilli, one bottle (65ml) daily (under supervision of a Health Worker) for 12 weeks and the control arm will receive a similar drink without the lactobacilli (Nutrient drink) daily for 12 weeks. Randomization will be done in a ratio of 1:1, i.e., the study arm and control arm will include 2000 children each. All the children under the study will be visited daily by a health worker who will supervise intake of Probiotic drink or Nutrient drink by the children. All the children will be followed up daily for 24weeks for identification of acute diarrhoea cases.

METHODOLOGY

Slum areas in Kolkata Municipal Corporation with approximately 60,000 populations (approximate 15,000 families) will be selected from ward 66 to reach a sample size of minimum 4,000 children (1-5 year age).

Baseline anthropometric measurements will be taken. The diarrhoeal surveillance will be through regular household visit by CHW and stool container will be kept at each child's house to collect stool sample if diarrhoea occurs.

INCLUSION/ EXCLUSION CRITERION FOR RECRUITMENT OF PARTICIPANTS Children of either sex aged 1-5 years will be eligible for screening and parents will give and a written, informed consent form (Appendix 7) will be required from either of the parents/ guardians of each participating child. Participating children should be free from any chronic illness and also any recent illness that may compromise the immune system. In general they will have good health without known underlying illness.

Children with history of diarrhoea in the preceding 2 weeks will not be eligible.

ADMINISTRATION OF STUDY AGENTS

There will be a setup of 5 health outposts and 20 clusters (each cluster with 40 children) will be approximately of 800 children will be assigned for each health outpost. There will be 20 Community Health Workers (CHW), allocated in each health outpost will be responsible for administer of one agent code for 40 children.

SAFETY EVALUATION

Clinical monitor will evaluate adverse events due to intake of the drink.

DATA MANAGEMENT PROCEDURES

Data obtained from demographic survey (Appendix 4), daily reports and other proforma will be entered in a PC using suitable software. Data will be scrutinized for accuracy and consistency before it is entered into the PC. Data will be entered into computers in a dedicated area located at NICED, using data entry programs specially created for the project by programmer.

STATISTICAL CONSIDERATIONS

Endpoints

Efficacy will be assessed by comparing the following between the probiotic and nutrient groups:

i) Average duration of diarrhoea ii) Severity of the disease iii) Incidence of diarrhoeal disease iv) Nutritional gain v) Analysis of fecal microflora

ETHICAL ASSURANCE FOR PROTECTION OF HUMAN RIGHTS

Written informed consent will be obtained from the parent/guardian of each participating child for the Probiotic and Nutrition studies and for the safety and for permission to collect feces. The probiotic or nutritional drink is safe and has been administered to infant children, adults and the elderly.

Storage conditions

The probiotic and nutrient will be stored at 4 to 10C. Bottles taken to the field will be carried in carrying bags. Each box will have a single ice pack, and care will be taken not to freeze the contents of the bottle.

MONITORING, AUDITING, INSPECTION

Responsibilities of the investigator(s)

The principal and co-investigators at NICED will be responsible for overall supervision and management of the project. Field investigators and other co-investigators will support the PI. The PI and co-investigators will supervise all activities at health facilities and in the sites (demographic surveillance, data collection, and samples collection and transportation). They will also visit the study sites regularly.

ETHICAL AND REGULATORY STANDARDS

Ethical principle

The justification for using a nutrient in this study is that: 1) no probiotic is currently recommended for use for prevention of diarrhoeal diseases in public health programs in India and 2) a valid assessment of probiotic efficacy in Kolkata, which is endemic for diarrhoea, can only be obtained with use of a nutrient. The nutrient will consist of nutrient without lactobacillus, which will help for nutritional growth of the children.

Potential benefits

During both phases of the project, the potential benefits to participants include proper treatment and referral when needed, as well as free and accurate diagnosis of the causative agent of diarrhoeal disease. During the trial phase, the probiotic recipients are expected to benefit from the protection offered by the probiotic against diarrhoea.

Potential risks

The potential risk to the participants will be minimal, since there is extensive documentation for the safety of the probiotic to be used.

Risk/benefit ratio

The direct benefit the participants may expect from participating in this study will be free laboratory examination and treatment for diarrhoea diseases.

The main benefit of obtaining data on the efficacy of the probiotic in Kolkata will be that these data will be crucial in guiding the decision of the Indian, and perhaps other developing country governments as to whether this probiotic will be alternative approach for growth of the children as well as prevention of diarrhoeal diseases. All recipients of the probiotic will potentially benefit from the probable protective effects against diarrhoea. The risks associated with the use of the probiotic or the nutrient and various other study procedures proposed to be used in this trial are expected to be minimal to nonexistent.

Laws and regulations

The study will be performed in accordance with the principles that govern biomedical research involving human subjects, specifically the ICMR Ethical Guidelines, the Declaration of Helsinki, and the International Conference on Harmonization's Good Clinical Practice Guidelines to provide assurance that the rights, integrity, and confidentiality of trial subjects are protected and that reported results are credible and accurate.

Informed consent

Individual informed consents from parents of eligible children between 1-5 years old will be obtained. Consent will be documented by signature or thumbprint of the parents/guardian on separate sheet. The privacy and confidentiality of all data and information collected from trial participants will be ensured both during and after the conduct of the trial. Individuals will not be identified in any reports and publications based on the trial data.

Institutional review committee

Before initiation of the study, the final protocol and the informed consent will require clearance Scientific Advisory Committee of NICED, Institutional Ethics Committee of NICED, Health Ministry Screening Committee of the Government of India.

ADMINISTRATIVE ASPECTS

Record retention

The principal investigator and NICED will keep all trial documents for at least 5 years after the completion or discontinuation of the study.

KEY PERSONNEL Name Professional Discipline/ Specialty Role in the Project

1. 1. Dipika Sur Epidemiology PI in India
2. 2. S.K. Bhattacharya Cholera and enteric disease Co-PI in India
3. 4. Byomkesh Manna Epidemiology Co-I in India
4. 5. S.K. Niyogi Microbiology Co-I in India
5. 6 Anup Palit Microbiology Co-I in India
6. 7. S.P. Mukhopadhyay Public health Controller
7. 8. Ashok Chowdhury Clinician Clinical Monitor

ELIGIBILITY:
Inclusion Criteria:

* Children of either sex aged 1-5 years will be eligible for screening and parents will give and a written, informed consent form will be required from either of the parents/ guardians of each participating child.
* Participating children should be free from any chronic illness and also any recent illness that may compromise the immune system. In general they will have good health without known underlying illness

Exclusion Criteria:

* Children below -2SD of the National Center for Health Statistics (NCHS) reference median in the nutritional parameters will not be enrolled.
* Children with history of diarrhoea in the preceding 2 weeks will not be eligible.

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4000 (Actual)
Dates: Start 2007-06; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Diarrhoeal episodes in children | 10 months

SECONDARY OUTCOMES:
nutritional status in children | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Dipika Sur, MD, Principal Investigator — National Institute of Cholera and Enteric Diseases, India
Locations (1):
- National Institute of Cholera and Enteric Disease, Kolkata, West Bengal, India

REFERENCES:
- [Derived] Sur D, Manna B, Niyogi SK, Ramamurthy T, Palit A, Nomoto K, Takahashi T, Shima T, Tsuji H, Kurakawa T, Takeda Y, Nair GB, Bhattacharya SK. Role of probiotic in preventing acute diarrhoea in children: a community-based, randomized, double-blind placebo-controlled field trial in an urban slum. Epidemiol Infect. 2011 Jun;139(6):919-26. doi: 10.1017/S0950268810001780. Epub 2010 Jul 30. PMID 20670468